CLINICAL TRIAL: NCT04621513
Title: Establishing the Collaborative Care Model of Traditional Chinse Medicine and Western Medicine for Allergic Rhinitis With Obstructive Sleep Apnea From Prevention to Treatment.
Brief Title: Collaborative Care Model for Allergic Rhinitis With Obstructive Sleep Apnea From Prevention to Treatment.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Wan-Yu Lai, Director, Division of Chinese Medicine Pediatrics, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH109-REC1-089
Record Dates: First submitted 2020-07-29; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Pediatric Sleep Apnea
MeSH Terms: interventions — montelukast

STUDY DESIGN:
Intervention Model Description: Parallel Randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative Care Model of TCM and WM (Experimental): Traditional Chinese Medicine(TCM):laser acupuncture and massage education. Western Medicine (WM):intra-nasal corticosteroid with singulair
  Interventions: Device: laser acupuncture (RJ laser S/N 1813458); Drug: western medicine
- Western medicine (Active Comparator): Western Medicine (WM):intra-nasal corticosteroid with singulair
  Interventions: Drug: western medicine

INTERVENTIONS:
Device: laser acupuncture (RJ laser S/N 1813458) — use a low-level-laser acupuncture on acupoint
  Arms: Collaborative Care Model of TCM and WM
Drug: western medicine — Montelukast 4mg 1 tablet HS AVAMYS nasal spray 27.5μg QD
  Other Names: intra-nasal corticosteroid(AVAMYS) with Montelukast (singulair)

SUMMARY:
In this project,the investigators aim to establish a Collaborative Care Model of TCM and Western Medicine to improve the quality of life and symptoms of AR with OSA children and educate care-givers diet and massage information to improve self-care ability and alleviate anxiety for parents. In addition, the investigators will use portable oxymeter to detect the change of SpO2 and respiratory arousal index daily at home and evaluate sensitivity and specificity of portable oxymeter device applied in OSA. The investigators want to give holistic health care for participants and care-givers by this project. In addition, the investigators will build a training environment to provide medical education and training opportunity to teach medical students and clinician the knowledge of pediatric allergic rhinitis and obstructive sleep apnea by caring patients and learning from clinical cases.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) affects 1-6% among children and has negative influence on day-time school performance and quality of sleep. It also cause failure to thrive，cardiovascular disease，and metabolic disease, which need early intervention. About 6% allergic rhinitis (AR) children would combine with OSA and refractory to treatment and need long-term intra-nasal corticosteroid or surgery if have moderate-severe OSA with adenoid-tonsillar hypertrophy. Some parents considering the side effect of steroid and risk of surgery will search Traditional Chinese Medicine (TCM) for help.

TCM is one kind of preventive medicine by educating people how to keep health by diet and massage. The breathing technique and "Teeth-Buckling and Salivary-Swallowing motion" noted in Inner Canon of the Yellow Emperor, one of the most important ancient Chinese medical text are compatible with myofunctional therapy for OSA. There are several studies revealed improve immune response in allergic rhinitis by TCM and severity of OSA by acupuncture.

In this project, the investigators aim to establish a Collaborative Care Model of TCM and Western Medicine to improve the quality of life and symptoms of AR with OSA children and educate care-givers diet and massage information to improve self-care ability and alleviate anxiety for parents. In addition, the investigators will use portable oxymeter to detect the change of SpO2 and respiratory arousal index daily at home and evaluate sensitivity and specificity of portable oxymeter device applied in OSA. The investigators want to give holistic health care for patients and care-givers by this project. In addition, the investigators will build a training environment to provide medical education and training opportunity to teach medical students and clinician the knowledge of pediatric allergic rhinitis and obstructive sleep apnea by caring patients and learning from clinical cases.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than 18 years old
2. Patients with persistent, moderate to severe allergic rhinitis who have been diagnosed by ARIA (2014) diagnostic criteria
3. AHI by polysomnography is >1 and diagnosis with obstructive sleep apnea.

Exclusion Criteria:

1. Abnormal craniofacial structure and require surgery.
2. Patients with sleep apnea caused by muscular dysplasia of the upper respiratory tract ( eg. cerebral palsy, Down syndrome, and other congenital muscular hypoplasia).
3. Mental or behavioral abnormalities that cannot cooperate with the researcher, such as schizophrenia, depression, suicidal ideation, etc.
4. Allergy to the treatment previously
5. Any disease or organ system dysfunction that may be life-threatening

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-12-16 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of mean score of Obstructive Sleep Apnea-18 Questionnaire | 8 weeks
  Evaluation quality of life pediatric Obstructive Sleep Apnea-18 ,(score:0-108)

SECONDARY OUTCOMES:
The change of mean score of Sinus and Nasal Quality of Life Survey | 8 weeks
  questionnaire for quality of life Sinus and Nasal disease (score:5-45)
The change of mean score of Pediatric Sleep Questionnaire | 8 weeks
  For quality of sleep (score:0-22)
The change of mean score of SNAP IV ( Swanson, Nolan and Pelham questionnaire) | 8 weeks
  for hyperactivity -tention deficiency disease (score:0-78)
Apnea-Hypopnea Index | 8 weeks
  by polysomnography
adeonid nasopharnygeal ratio | 8 weeks
  by X ray Cephalometry
tonsil size | 8 weeks
  Friedman Grading Scale (grade 0-4)
nasal volume | 8 weeks AND 12 weeks
  Acoustic rhinometry
adenoid size | 8 weeks
  Clemen and McMurray grade 1-4

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University & Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No